CLINICAL TRIAL: NCT03717701
Title: Combining Metformin and Esomeprazole in Treatment of Early Onset Preeclampsia: A Double-Blind Randomized, Placebo-controlled Trial
Brief Title: Metformin and Esomeprazole in Treatment of Early Onset Preeclampsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: aswu/273/9l18
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Pre-Eclampsia
Keywords: preeclampsia; esomeprazole; metformin
MeSH Terms: conditions — Pre-Eclampsia | interventions — Metformin; Esomeprazole

STUDY DESIGN:
Intervention Model Description: This is a randomized double-blinded placebo-controlled intervention trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: both participants and researchers will be blinded to the intervention given
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- metformin and esomeprazole (Experimental): Patients will take esomeprazole single dose of 40 mg orally once a day plus single dose of metformin 1000mg orally single dose once a day
  Interventions: Drug: metformin; Drug: esomeprazole
- Placebo (Placebo Comparator): Patients will take inert tablets similar in appearance, color, and consistency
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: metformin — Patients will take metformin single dose of 1000 mg orally once a day
  Other Names: Experimental
  Arms: metformin and esomeprazole
Drug: esomeprazole — Patients will take esomeprazole single dose of 40 mg orally once a day
  Other Names: Experimental
  Arms: metformin and esomeprazole
Drug: Placebo — Patients will take inert tablets similar in appearance, color, and consistency
  Arms: Placebo

SUMMARY:
Preeclampsia is globally responsible for tens of thousands of maternal and neonatal deaths each year. Currently, there are no medical therapies to halt disease progression and expectant management and delivery remain the mainstay of treatment. An important step in the pathogenesis of preeclampsia is a poor placental invasion and the subsequent release of the anti-angiogenic factors soluble fms-like tyrosine kinase 1 (sFlt-1) and soluble endoglin (sEng)into the maternal circulation. Given metformin and esomeprazole successfully mitigate key pathogenic features of preeclampsia, the investigator will study whether combining low-doses of metformin and esomeprazole may be additive or synergistic (or neither) in reducing sFlt-1 and sEng secretion, and mitigating endothelial dysfunction, compared to placebo.

DETAILED DESCRIPTION:
This is a randomized double-blinded placebo-controlled intervention trial investigating preeclampsia, defined according to the International Society for the Study of Hypertension in Pregnancy (ISSHP). The population of interest involves pregnant women diagnosed with pre-eclampsia at a gestational age between 28 and 32 weeks at Aswan university hospital will be invited to participate. To be enrolled, the treating team needs to have determined after their initial assessment that delivery is unlikely to be required within 48 h. A starting point of 28 weeks has been chosen as this would be the earliest gestation that Aswan university hospital to be viable and are suitable to be offered expectant management The intervention involves randomization to oral esomeprazole tablets40 mg plus metformin tablets 1000 mg or identical placebo tablets from recruitment until delivery. Randomization is achieved using computational random allocation, and both participants and researchers will be blinded to the intervention given.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women presenting at a Gestational age between 28 + 0 weeks and 32 + 0 weeks presented with preterm preeclampsia
* The patient will be managed with an expectant management
* Give written informed consent

Exclusion Criteria:

* Multiple pregnancies.
* Previous hypersensitivity reaction esomeprazole or metformin
* Contraindications to the use of esomeprazole or metformin
* The patient is unable or unwilling to give consent
* An established fetal compromise that necessitates delivery
* The presence of any of the following at presentation:

  * Eclampsia.
  * Severe hypertension.
  * A cerebrovascular event as an ischemic or hemorrhagic stroke.
  * Renal impairment.
  * Signs of left ventricular failure which include pulmonary edema.
  * Disseminated intravascular coagulation (DIC)
  * Haemolysis, elevated liver enzymes and low platelets (HELLP syndrome)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women with early-onset preeclampsia
Enrollment: 120 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Prolongation of gestation measured from the time of enrollment to the time of delivery. | 4 weeks
  Prolongation of gestation measured from the time of enrollment to the time of delivery.

SECONDARY OUTCOMES:
Severe morbidity | 4 weeks
  Severe morbidity including eclampsia, liver or renal failure, hemolysis, elevated liver enzymes and low platelets syndrome (HELLP), disseminated intravascular coagulation (DIC), stroke, and pulmonary edema
The change in serum level of sFlt-1 and endoglin before the start of treatment and at termination of pregnancy | 4 weeks
  The change in serum level of sFlt-1 and endoglin before the start of treatment and at termination of pregnancy
Side effects | 4 weeks
  any side effects or adverse events related to the intervention, intervention stopped due to side effects

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No